CLINICAL TRIAL: NCT02880852
Title: A Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK1550188 in Chinese Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Belimumab Phase I Study in Chinese Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200909
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Belimumab; Pharmacodynamics; safety tolerability; Pharmacokinetics; Chinese subjects
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belimumab 10 mg/kg (Experimental): In this open label study, a single dose of 10 mg/kg Belimumab will be administered intravenously in Chinese subjects with systemic lupus erythematosus.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab will be provided as white uniform lyophilized cake in vials with unit dose strength of 400 mg/vial plus excipients (citric acid/sodium citrate/sucrose/polysorbate) for reconstitution in 4.8 milliliter sterile water for injection (SWFI). Belimumab will be administered as 10 mg/kg intravenous infusion for over 1 hour on Day 0.

SUMMARY:
In China, Belimumab (GSK1550188) will be developed for a dosing regimen of once-monthly intravenous (IV) infusion for the treatment of SLE. This open-label, single dose study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of belimumab in Chinese SLE subjects. A total of approximately 20 subjects will be enrolled to receive IV infusion of 10 milligrams per kilogram (mg/kg) GSK1550188 on Day 0 for the treatment of SLE. Subjects will be followed for 84 days after the administration of drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who give consent to this study participation and sign informed consent form.
* Subjects at least 18 years of age inclusive at screening visit.
* SLE Classification: Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) classification criteria, with 4 or more of the 11 ACR criteria present, serially or simultaneously during any interval or observation.
* SLE Treatment: Be on either no SLE medication or a stable SLE treatment regimen of any medication (alone or in combination) for a period of at least 2 months prior to Day 0; corticosteroids (prednisone or prednisone equivalent, up to 40 mg/day); immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium), mizoribine, calcineurin inhibitors (example [e.g.], tacrolimus, cyclosporine), sirolimus, oral cyclophosphamide, 6-mercaptopurine, or thalidomide; anti-malarials (e.g., hydroxychloroquine, chloroquine, quinacrine) and non-steroidal anti-inflammatory drugs (NSAIDs).
* The subjects with positive test for anti-nuclear antibody (ANA) or anti-double stranded deoxyribonucleic acid (DNA) serum antibody.
* Males and females: A female subject is eligible to enter the study if she is: not pregnant or nursing; of non-childbearing potential (i.e., women who had a hysterectomy, are postmenopausal which is defined as 1 year without menses, have both ovaries surgically removed or have current documented tubal ligation); of childbearing potential (i.e., women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea [even severe], women who are perimenopausal or have just begun to menstruate. These women must have a negative serum pregnancy test at screening, and agree to one of the following: complete abstinence from penile-vaginal intercourse, when this is the female's preferred and usual lifestyle, from 2 weeks prior to administration of the 1st dose of investigational product (IP) until study complete; or consistent and correct use of one of the following acceptable methods of birth control for 1 month prior to the start of the IP and for 16 weeks after the last dose of IP: any intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1 percent (%) per year; oral contraceptives; double barrier method with vaginal spermicidal agent: condom and an occlusive cap (cervical cap/vault or diaphragm) with a vaginal spermicidal agent (foam/gel/film/cream/suppository); implants of etonogestrel or levonorgestrel; estrogenic vaginal ring; injectable progesterone; percutaneous contraceptive patch; male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subject.
* Based on single or averaged corrected QT (QTc) interval values of triplicate ECGs obtained over a brief recording period: [QTc corrected by Bazett's (QTcB) or QTc corrected by Fridericia's (QTcF) formula] <450 milliseconds (msec); or QTcB or QTcF <480 msec in subjects with bundle branch block.

Exclusion Criteria:

* B-cell Therapy: Have received treatment with any B cell targeted therapy (e.g., rituximab, other anti-CD20 agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], Transmembrane activator and calcium-modulator and cytophilin ligand interactor [TACI] Fc, or belimumab) at any time.
* The subject has received a biologic investigational or non-investigational agent within 12 months prior to Day 0.
* Received IV immunoglobulin (Ig), plasmapheresis, hemodialysis, intravenous cyclophosphamide, or high dose prednisone and its equivalents (>60 mg/day) within 6 months prior to Day 0.
* The subject has received a non-biologic investigational agent within 2 months prior to Day 0.
* The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational agent.
* The subject has severe lupus kidney disease (defined by proteinuria >6 grams [g]/24 hours) within 6 months prior to the Screening visit.
* History of renal transplant.
* Active central nervous system (CNS) lupus [including seizures, psychosis, organic brain syndrome, cerebrovascular accident (CVA), motor neuropathy, vasculitis] requiring medical intervention within 6 months prior to Screening visit.
* Infections: Have required management of acute or chronic infections, as follows: currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria); hospitalization for treatment of infection within 2 months prior to Day 0; use of parenteral (IV or intramuscular [IM]) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 2 months prior to Day 0.
* The subject has hypogammaglobulinemia or immunoglobulin A (IgA) deficiency (IgA level <10 mg/deciliter [dL]).
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Uncontrolled other diseases: History or clinical evidence of active significant acute or chronic diseases (i.e., cardiovascular, pulmonary, untreated hypertension, anemia, gastrointestinal, hepatic, renal, neurological, cancer, or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* Have a planned surgical procedure, or a history of any other medical disease, or laboratory abnormalities, or conditions which would make the subject (in the opinion of the Investigator) unsuitable for the study.
* The subject has an abnormality on 12-lead ECG at screening which is clinically significant in the opinion of the investigator.
* Have evidence of current drug or alcohol abuse or dependence.
* AST and ALT >=2x upper limit of normal (ULN); ALP and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Have a historically positive human immunodeficiency virus (HIV) test or test positive at screening for HIV.
* History of or positive test at screening visit for any of Hepatitis B surface antigen (HBsAg), anti- Hepatitis B core antibody (HBcAb) or anti-hepatitis C virus antibodies (HCVAb). If only anti-HBcAb result is positive, hepatitis B virus (HBV)-(DNA) test will be performed. If HBV-DNA results in negative, the patient is eligible.
* Laboratory Abnormalities: Have a Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:
* Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
* Stable Grade 3/4 proteinuria (=<6 g/24 hour equivalent by spot urine protein to creatinine ratio allowed).
* Stable Grade 3 hypoalbuminemia due to lupus nephritis, and not related to liver disease or malnutrition.
* Stable Grade 3 neutropenia or stable Grade 3 white blood cell count.
* Subjects who have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months or who, in the investigator's opinion, pose a significant suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20304

REFERENCES:
- [Background] Zhang J, Wan W, Miao L, Wu J, Dong J, Shen Y, Xiong C, Li C, Xue Y, Cao G, Ma P. Pharmacokinetics, Pharmacodynamics and Safety of Belimumab in Chinese Patients with Systemic Lupus Erythematosus: A Phase I, Open-Label Study. Rheumatol Ther. 2020 Mar;7(1):191-200. doi: 10.1007/s40744-020-00193-9. Epub 2020 Jan 17. PMID 31953740
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants with Systemic Lupus Erythematosus (SLE) were enrolled. The study was conducted at 2 centers in China from 23-Jan-2017 to 08-Sep-2017.
Pre-assignment Details: A total of 25 participants were screened, of which 5 participants were screen failures. The reason for screen failures were: did not meet inclusion/exclusion criteria (4 participants) and investigator discretion (1 participant).
Groups:
- Belimumab 10 mg/kg: Eligible participants received a single dose of belimumab 10 milligrams (mg) per kilogram (kg) as intravenous infusion for over an hour on Day 0.
Period: Overall Study
Arm/Group | Belimumab 10 mg/kg
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population which comprised of all the participants who received at least one dose of study medication.
Groups:
- Belimumab 10 mg/kg: Eligible participants received a single dose of belimumab 10 mg per kg as intravenous infusion for over an hour on Day 0.
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Belimumab
Description: Blood samples were collected at the indicated timepoints to calculate Cmax of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: Pharmacokinetic (PK) Parameter Population, which comprised of all those participants who received a dose of belimumab and for whom PK parameters could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Micrograms per milliliter | 221.3532 (12.8405)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0 to t]) and Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0 to Inf]) of Belimumab
Description: Blood samples were collected at the indicated timepoints to calculate AUC (0 to t) and AUC (0 to inf) of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms/milliliter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Day*micrograms/milliliter
  AUC(0 to t) | 2395.3030 (23.2924)
  AUC(0 to inf) | 2461.8013 (24.7125)

3. Primary Outcome: Terminal Phase Half-life (t1/2) of Belimumab
Description: Blood samples were collected at the indicated time points to calculate t1/2 of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Days | 14.6283 (35.4339)

4. Primary Outcome: Terminal Phase Rate Constant (Lambda z) of Belimumab
Description: Blood samples were collected at the indicated time points to calculate lambda z of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/day
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
1/day | 0.0474 (35.4339)

5. Primary Outcome: Systemic Clearance (CL) of Belimumab
Description: Blood samples were collected at the indicated time points to calculate CL of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (Milliliters/day)/kilogram
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
(Milliliters/day)/kilogram | 4.0621 (24.7125)

6. Primary Outcome: Volume of Distribution (Vz) of Belimumab
Description: Blood samples were collected at the indicated time points to calculate Vz of belimumab.
Time Frame: Day 0 (pre-dose, 5 minutes, 1 hour, 6 hours, 24 hours), and on Days 1, 7, 14, 21, 28, 42, 56, and 84 post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters/kilogram
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Milliliters/kilogram | 85.7265 (21.6704)

7. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant, or associated with liver injury and impaired liver function.
Time Frame: Up to Day 84
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Participants
  AE | 12
  SAE | 1

8. Secondary Outcome: Change From Baseline to Day 84 in Vital Signs- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs included SBP and DBP. SBP and DBP were measured with the participant in the sitting position. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Millimeters of mercury
  DBP: Day 0 (5 minutes post-dose) | -0.5 (6.35)
  DBP: Day 0 (1 hour post-dose) | -1.5 (12.51)
  DBP: Day 0 (6 hours post-dose) | -2.1 (8.57)
  DBP: Day 0 (24 hours post-dose) | -0.1 (7.95)
  DBP: Day 1 | 2.2 (8.37)
  DBP: Day 7 | 1.1 (7.91)
  DBP: Day 14 | 0.5 (8.65)
  DBP: Day 21 | 0.1 (6.91)
  DBP: Day 28 | 0.2 (8.86)
  DBP: Day 42 | -3.2 (7.99)
  DBP: Day 56 | -0.8 (8.85)
  DBP: Day 84 | -0.6 (11.06)
  SBP: Day 0 (5 minutes post-dose) | 0.8 (9.92)
  SBP: Day 0 (1 hour post-dose) | -2.5 (11.44)
  SBP: Day 0 (6 hours post-dose) | -4.5 (12.15)
  SBP: Day 0 (24 hours post-dose) | -3.7 (11.76)
  SBP: Day 1 | -2.4 (10.92)
  SBP: Day 7 | 0.7 (10.65)
  SBP: Day 14 | -1.0 (12.09)
  SBP: Day 21 | -4.4 (12.05)
  SBP: Day 28 | -1.5 (14.01)
  SBP: Day 42 | -7.4 (9.26)
  SBP: Day 56 | -4.0 (11.14)
  SBP: Day 84 | -7.4 (14.91)

9. Secondary Outcome: Change From Baseline to Day 84 in Vital Sign- Pulse Rate
Description: Vital signs included pulse rate. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Beats per minute
  Day 0 (5 minutes post-dose) | -1.2 (11.13)
  Day 0 (1 hour post-dose) | -1.6 (8.43)
  Day 0 (6 hours post-dose) | 2.6 (12.14)
  Day 0 (24 hours post-dose) | 2.3 (11.08)
  Day 1 | 5.7 (11.09)
  Day 7 | 4.7 (11.82)
  Day 14 | 6.9 (10.55)
  Day 21 | 5.0 (8.90)
  Day 28 | 7.6 (10.02)
  Day 42 | 8.3 (12.06)
  Day 56 | 4.1 (10.80)
  Day 84 | 3.2 (14.21)

10. Secondary Outcome: Change From Baseline to Day 84 in Vital Sign- Temperature
Description: Vital signs included temperature. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Celsius
  Day 0 (5 minutes post-dose) | 0.21 (0.485)
  Day 0 (1 hour post-dose) | 0.17 (0.473)
  Day 0 (6 hours post-dose) | 0.20 (0.552)
  Day 0 (24 hours post-dose) | 0.40 (0.617)
  Day 1 | 0.24 (0.486)
  Day 7 | 0.40 (0.793)
  Day 14 | 0.40 (0.504)
  Day 21 | 0.41 (0.454)
  Day 28 | 0.37 (0.457)
  Day 42 | 0.53 (0.595)
  Day 56 | 0.52 (0.473)
  Day 84 | 0.38 (0.434)

11. Secondary Outcome: Number of Participants With Abnormal-clinically Significant 12-lead Electrocardiogram (ECG) Findings
Description: ECG parameters included heart rate, PR interval, QRS interval, QT interval and corrected QT (QTc) interval. Number of participants with abnormal-clinically significant 12-lead ECG findings are presented.
Time Frame: Up to Day 84
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Participants | 0

12. Secondary Outcome: Change From Baseline to Day 84 in Clinical Chemistry Parameters- Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase
Description: Clinical chemistry parameters included ALT, ALP, AST, GGT and lactate dehydrogenase. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
International units per Liter (IU/L)
  ALT: Day 0 (24 hours) | -1.6 (3.46)
  ALT: Day 14 | -1.3 (11.93)
  ALT: Day 28 | -3.2 (12.34)
  ALT: Day 56 | -5.0 (12.18)
  ALT: Day 84 | -5.5 (11.84)
  ALP: Day 0 (24 hours) | -3.9 (3.56)
  ALP: Day 14 | -5.6 (10.72)
  ALP: Day 28 | -3.4 (8.80)
  ALP: Day 56 | -7.2 (9.26)
  ALP: Day 84 | -7.3 (11.80)
  AST: Day 0 (24 hours) | -1.9 (2.48)
  AST: Day 14 | -1.8 (8.58)
  AST: Day 28 | -2.6 (8.46)
  AST: Day 56 | -2.8 (6.15)
  AST: Day 84 | -3.6 (6.86)
  GGT: Day 0 (24 hours) | -1.5 (2.33)
  GGT: Day 14 | -0.5 (7.34)
  GGT: Day 28 | 0.5 (7.22)
  GGT: Day 56 | -4.1 (6.08)
  GGT: Day 84 | -3.3 (8.44)
  Lactate dehydrogenase: Day 0 (24 hours) | -8.1 (10.56)
  Lactate dehydrogenase: Day 14 | -3.2 (18.88)
  Lactate dehydrogenase: Day 28 | -1.4 (22.30)
  Lactate dehydrogenase: Day 56 | 1.3 (24.30)
  Lactate dehydrogenase: Day 84 | 1.5 (20.68)

13. Secondary Outcome: Change From Baseline to Day 84 in Clinical Chemistry Parameters- Albumin and Protein
Description: Clinical chemistry parameters included albumin and protein. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Grams per liter (g/L)
  Albumin: Day 0 (24 hours) | -1.4 (1.88)
  Albumin: Day 14 | -1.1 (3.08)
  Albumin: Day 28 | -0.6 (2.68)
  Albumin: Day 56 | -0.5 (3.14)
  Albumin: Day 84 | -0.6 (3.10)
  Protein: Day 0 (24 hours) | -3.8 (2.67)
  Protein: Day 14 | -3.2 (5.12)
  Protein: Day 28 | -3.3 (4.47)
  Protein: Day 56 | -3.8 (5.41)
  Protein: Day 84 | -3.8 (4.23)

14. Secondary Outcome: Change From Baseline to Day 84 in Clinical Chemistry Parameters- Bilirubin, Creatinine, Direct Bilirubin, Indirect Bilirubin and Urate
Description: Clinical chemistry parameters included bilirubin, creatinine, direct bilirubin, indirect bilirubin and urate. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (µmol/L)
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Micromoles per Liter (µmol/L)
  Bilirubin: Day 0 (24 hours) | -2.8 (3.07)
  Bilirubin: Day 14 | -2.4 (4.48)
  Bilirubin: Day 28 | -3.4 (4.55)
  Bilirubin: Day 56 | -3.2 (5.17)
  Bilirubin: Day 84 | -2.1 (4.83)
  Creatinine: Day 0 (24 hours) | -0.18 (4.479)
  Creatinine: Day 14 | -0.80 (5.502)
  Creatinine: Day 28 | -0.43 (6.698)
  Creatinine: Day 56 | -0.25 (5.962)
  Creatinine: Day 84 | -0.18 (6.062)
  Direct bilirubin: Day 0 (24 hours) | -0.4 (1.05)
  Direct bilirubin: Day 14 | 0.1 (1.37)
  Direct bilirubin: Day 28 | -0.6 (1.14)
  Direct bilirubin: Day 56 | -0.6 (1.47)
  Direct bilirubin: Day 84 | -0.2 (1.28)
  Indirect bilirubin: Day 0 (24 hours) | -2.4 (2.87)
  Indirect bilirubin: Day 14 | -2.5 (4.10)
  Indirect bilirubin: Day 28 | -2.8 (4.12)
  Indirect bilirubin: Day 56 | -2.6 (4.26)
  Indirect bilirubin: Day 84 | -1.9 (4.79)
  Urate: Day 0 (24 hours) | -14.5 (21.88)
  Urate: Day 14 | -10.5 (34.41)
  Urate: Day 28 | -13.5 (47.49)
  Urate: Day 56 | -2.5 (49.93)
  Urate: Day 84 | -7.5 (50.67)

15. Secondary Outcome: Change From Baseline to Day 84 in Clinical Chemistry Parameters- Calcium, Calcium Corrected, Carbon Dioxide, Chloride, Magnesium, Phosphate, Potassium, Sodium, Urea and Glucose
Description: Clinical chemistry parameters included calcium, calcium corrected, carbon dioxide, chloride, magnesium, phosphate, potassium, sodium, urea and glucose. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Millimoles per Liter (mmol/L)
  Calcium: Day 0 (24 hours) | -0.040 (0.0599)
  Calcium: Day 14 | -0.020 (0.1049)
  Calcium: Day 28 | 0.004 (0.0848)
  Calcium: Day 56 | -0.020 (0.1054)
  Calcium: Day 84 | -0.027 (0.0909)
  Calcium Corrected: Day 0 (24 hours) | -0.010 (0.0466)
  Calcium Corrected: Day 14 | 0.003 (0.0663)
  Calcium Corrected: Day 28 | 0.017 (0.0578)
  Calcium Corrected: Day 56 | -0.007 (0.0694)
  Calcium Corrected: Day 84 | -0.016 (0.0501)
  Carbon dioxide: Day 0 (24 hours) | -0.3 (1.86)
  Carbon dioxide: Day 14 | -0.2 (2.32)
  Carbon dioxide: Day 28 | 0.1 (2.09)
  Carbon dioxide: Day 56 | -0.1 (2.33)
  Carbon dioxide: Day 84 | -0.2 (1.64)
  Chloride: Day 0 (24 hours) | 1.3 (2.12)
  Chloride: Day 14 | 0.3 (2.05)
  Chloride: Day 28 | 0.4 (1.53)
  Chloride: Day 56 | 1.3 (1.63)
  Chloride: Day 84 | 1.2 (1.74)
  Magnesium: Day 0 (24 hours) | -0.044 (0.0564)
  Magnesium: Day 14 | -0.046 (0.0623)
  Magnesium: Day 28 | -0.049 (0.0709)
  Magnesium: Day 56 | -0.029 (0.0750)
  Magnesium: Day 84 | -0.034 (0.0751)
  Phosphate: Day 0 (24 hours) | -0.085 (0.1299)
  Phosphate: Day 14 | -0.132 (0.2104)
  Phosphate: Day 28 | -0.135 (0.2201)
  Phosphate: Day 56 | -0.140 (0.2037)
  Phosphate: Day 84 | -0.152 (0.1509)
  Potassium: Day 0 (24 hours) | -0.10 (0.333)
  Potassium: Day 14 | -0.04 (0.355)
  Potassium: Day 28 | -0.11 (0.335)
  Potassium: Day 56 | -0.13 (0.370)
  Potassium: Day 84 | -0.29 (0.356)
  Sodium: Day 0 (24 hours) | 0.1 (2.24)
  Sodium: Day 14 | 0.3 (1.59)
  Sodium: Day 28 | 0.1 (1.28)
  Sodium: Day 56 | 0.8 (1.68)
  Sodium: Day 84 | 0.8 (1.67)
  Urea: Day 0 (24 hours) | 0.20 (0.733)
  Urea: Day 14 | 0.38 (1.122)
  Urea: Day 28 | 0.10 (1.382)
  Urea: Day 56 | -0.13 (0.793)
  Urea: Day 84 | -0.20 (1.152)
  Glucose: Day 0 (24 hours) | 0.98 (3.248)
  Glucose: Day 14 | 1.66 (2.094)
  Glucose: Day 28 | 0.33 (2.230)
  Glucose: Day 56 | 0.19 (2.093)
  Glucose: Day 84 | 0.57 (2.749)

16. Secondary Outcome: Change From Baseline to Day 84 in Hematology Laboratory Parameters- Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Hematology parameters included basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
10^9 cells/Liter
  Basophils: Day 0 (24 hours) | -0.006 (0.0110)
  Basophils: Day 14 | -0.011 (0.0176)
  Basophils: Day 28 | -0.013 (0.0186)
  Basophils: Day 56 | -0.008 (0.0162)
  Basophils: Day 84 | -0.005 (0.0115)
  Eosinophils: Day 0 (24 hours) | -0.019 (0.0506)
  Eosinophils: Day 14 | -0.024 (0.0564)
  Eosinophils: Day 28 | -0.006 (0.0535)
  Eosinophils: Day 56 | -0.022 (0.0595)
  Eosinophils: Day 84 | -0.028 (0.0670)
  Leukocytes: Day 0 (24 hours) | 0.29 (0.899)
  Leukocytes: Day 14 | 0.09 (1.403)
  Leukocytes: Day 28 | 1.00 (1.589)
  Leukocytes: Day 56 | 0.54 (1.337)
  Leukocytes: Day 84 | -0.04 (1.754)
  Lymphocytes: Day 0 (24 hours) | -0.068 (0.5214)
  Lymphocytes: Day 14 | -0.180 (0.6718)
  Lymphocytes: Day 28 | -0.364 (0.6746)
  Lymphocytes: Day 56 | -0.287 (0.5812)
  Lymphocytes: Day 84 | -0.257 (0.5697)
  Monocytes: Day 0 (24 hours) | 0.005 (0.1300)
  Monocytes: Day 14 | -0.025 (0.1575)
  Monocytes: Day 28 | -0.077 (0.2568)
  Monocytes: Day 56 | -0.076 (0.1574)
  Monocytes: Day 84 | -0.059 (0.1878)
  Neutrophils: Day 0 (24 hours) | 0.389 (0.9085)
  Neutrophils: Day 14 | 0.332 (1.8713)
  Neutrophils: Day 28 | 1.464 (1.9750)
  Neutrophils: Day 56 | 0.932 (1.3943)
  Neutrophils: Day 84 | 0.305 (1.7297)
  Platelets: Day 0 (24 hours) | -6.3 (12.68)
  Platelets: Day 14 | 2.1 (26.11)
  Platelets: Day 28 | 10.0 (30.14)
  Platelets: Day 56 | 1.0 (20.84)
  Platelets: Day 84 | -4.1 (29.04)

17. Secondary Outcome: Change From Baseline to Day 84 in Hematology Parameter- Erythrocytes
Description: Hematology parameter included erythrocytes. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
10^12 cells/Liter
  Day 0 (24 hours) | -0.12 (0.158)
  Day 14 | -0.19 (0.246)
  Day 28 | -0.13 (0.205)
  Day 56 | -0.16 (0.239)
  Day 84 | -0.18 (0.282)

18. Secondary Outcome: Change From Baseline to Day 84 in Hematology Parameter- Hematocrit
Description: Hematology parameter included hematocrit. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Proportion of red blood cells in blood
  Day 0 (24 hours) | -0.0112 (0.0170)
  Day 14 | -0.0176 (0.0272)
  Day 28 | 0.0006 (0.0310)
  Day 56 | -0.0060 (0.0226)
  Day 84 | -0.0126 (0.0313)

19. Secondary Outcome: Change From Baseline to Day 84 in Hematology Parameter- Hemoglobin
Description: Hematology parameter included hemoglobin. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Grams per Liter (g/L)
  Day 0 (24 hours) | -3.7 (4.83)
  Day 14 | -5.0 (7.14)
  Day 28 | -4.0 (5.55)
  Day 56 | -5.0 (8.04)
  Day 84 | -5.7 (10.11)

20. Secondary Outcome: Number of Participants With Positive Urinalysis Dipstick Results
Description: Urinalysis was done by the dipstick method to detect the presence of protein, glucose, ketones and occult blood in urine. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine occult blood, urine protein and urine ketones can be read as negative, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations in the urine sample; results for urinalysis parameter of urine glucose can be read as negative, Trace, 1+ or 1/4 gram per Liter (g/L), 2+ or 1/2 g/L, 3+ or 1 g/L and 4+ indicating proportional concentrations in the urine sample. *a indicates two participants did not take the urinalysis test at Day 14 on scheduled date but took an unscheduled sample at the next visit (Day 21) and *b indicates one participant did not take the urinalysis test at Day 28 on scheduled date but took an unscheduled sample at the next visit (Day 42). Only those participants with positive results have been presented.
Time Frame: Day 0 (24 hours), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 84
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Participants
  Glucose: Day 14, 1+ or 1/4 g/L | 1
  Glucose: Day 14, 2+ or 1/2 g/L | 1
  Glucose: Day 14, Trace | 1
  Glucose: Day 28, 1+ or 1/4 g/L | 1
  Glucose: Day 56, 1+ or 1/4 g/L | 1
  Occult Blood: Day 0 (24 hours), Trace | 5
  Occult Blood: Day 0 (24 hours), 1+ | 1
  Occult Blood: Day 0 (24 hours), 3+ | 1
  Occult Blood: Day 14, Trace | 4
  Occult Blood: Day 14, 1+ | 2
  Occult Blood: Day 14, 2+ | 1
  Occult Blood: Day 21*a, Trace | 1
  Occult Blood: Day 28, Trace | 6
  Occult Blood: Day 28, 2+ | 2
  Occult Blood: Day 56, Trace | 5
  Occult Blood: Day 56, 1+ | 2
  Occult Blood: Day 56, 2+ | 2
  Occult Blood: Day 84, Trace | 1
  Occult Blood: Day 84, 1+ | 3
  Occult Blood: Day 84, 2+ | 1
  Protein: Day 0 (24 hours), 2+ | 1
  Protein: Day 14, Trace | 3
  Protein: Day 14, 1+ | 1
  Protein: Day 28, 2+ | 1
  Protein: Day 42*b, Trace | 1
  Protein: Day 56, Trace | 2
  Protein: Day 84, Trace | 3
  Protein: Day 84, 2+ | 1

21. Secondary Outcome: Percent Change From Baseline to Day 84 in B Cell Subsets (Cluster of Differentiation [CD]19 and CD 20+) for Pharmacodynamic Assessment
Description: Immunoglobulin B cell subsets included CD19 and CD 20+. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value. Percent change from Baseline was calculated as 100 multiplied by [(Post-Baseline Visit Value minus Baseline) / Baseline]. Pharmacodynamic population comprised of participants who received the study medication and for whom pharmacodynamic data was available.
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed represented by n=X in the category titles.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Percent change
  CD19: Day 14, n=20 | 26.6444 (78.2275)
  CD19: Day 28, n=20 | -4.1141 (49.0574)
  CD19: Day 42, n=19: number analyzed (Participants) | 19
  CD19: Day 42, n=19 | -12.6852 (46.6312)
  CD19: Day 56, n=20 | -20.4908 (44.2536)
  CD19: Day 84, n=20 | -27.0912 (49.5965)
  CD20+: Day 14, n=20 | 35.3407 (100.7209)
  CD20+: Day 28, n=20 | 0.3444 (54.1435)
  CD20+: Day 42, n=19: number analyzed (Participants) | 19
  CD20+: Day 42, n=19 | -8.6327 (52.1804)
  CD20+: Day 56, n=20 | -20.6313 (42.8535)
  CD20+: Day 84, n=20 | -23.7421 (62.8031)

22. Secondary Outcome: Percent Change From Baseline to Day 84 in B Cell Subsets (CD20+/27+ Memory and CD20+/27-naïve) for the Pharmacodynamic Assessment
Description: Immunoglobulin B cell subset included CD20+/27+ memory and CD20+/27-naïve. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value. Percent change from Baseline was calculated as 100 multiplied by [(Post-Baseline Visit Value minus Baseline) / Baseline].
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Percent change
  CD20+/27+ memory: Day 14, n=20 | 186.4701 (199.5187)
  CD20+/27+ memory: Day 28, n=20 | 118.1433 (135.2351)
  CD20+/27+ memory: Day 42, n=19: number analyzed (Participants) | 19
  CD20+/27+ memory: Day 42, n=19 | 91.2965 (125.1803)
  CD20+/27+ memory: Day 56, n=20 | 135.8139 (167.0084)
  CD20+/27+ memory: Day 84, n=20 | 70.6332 (108.1058)
  CD20+/27-naïve: Day 14, n=20 | 4.0530 (61.8752)
  CD20+/27-naïve: Day 28, n=20 | -15.9190 (48.8363)
  CD20+/27-naïve: Day 42, n=19: number analyzed (Participants) | 19
  CD20+/27-naïve: Day 42, n=19 | -17.0090 (61.5514)
  CD20+/27-naïve: Day 56, n=20 | -40.2078 (37.1774)
  CD20+/27-naïve: Day 84, n=20 | -42.6608 (43.8690)

23. Secondary Outcome: Percent Change From Baseline to Day 84 in Immunoglobulins B Cell Subset (Normalized [Norm] CD19+/27BRIGHT[Br]/38Br SLE Subset, Norm CD20+/138+Plasmacytoid, Norm CD20+/69+Activated and Norm CD20-/CD138+Plasma Cell) for Pharmacodynamic Assessment
Description: Immunoglobulin B cell subset inlcuded Norm CD19+/27Br/38Br SLE subset, Norm CD20+/138+plasmacytoid, Norm CD20+/69+activated and Norm CD20-/CD138+plasma cell. Baseline was pre-dose on Day 0. Change from Baseline was defined as the post-Baseline value minus the Baseline value. Percent change from Baseline was calculated as 100 multiplied by [(Post-Baseline Visit Value minus Baseline) / Baseline].
Time Frame: Baseline (pre-dose on Day 0) to Day 84
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 20
Percent change
  Norm CD19+/27Br/38Br SLE subset: Day 14, n=20 | 5.3271 (85.7472)
  Norm CD19+/27Br/38Br SLE subset: Day 28, n=20 | -4.4623 (91.3321)
  Norm CD19+/27Br/38Br SLE subset: Day 42, n=19: number analyzed (Participants) | 19
  Norm CD19+/27Br/38Br SLE subset: Day 42, n=19 | 17.2492 (132.2146)
  Norm CD19+/27Br/38Br SLE subset: Day 56, n=20 | 48.1481 (148.1877)
  Norm CD19+/27Br/38Br SLE subset: Day 84, n=20 | 24.9838 (118.1567)
  Norm CD20+/138+plasmacytoid: Day 14, n=19: number analyzed (Participants) | 19
  Norm CD20+/138+plasmacytoid: Day 14, n=19 | 200.6464 (702.0072)
  Norm CD20+/138+plasmacytoid: Day 28, n=19: number analyzed (Participants) | 19
  Norm CD20+/138+plasmacytoid: Day 28, n=19 | 255.8559 (1010.9303)
  Norm CD20+/138+plasmacytoid: Day 42, n=18: number analyzed (Participants) | 18
  Norm CD20+/138+plasmacytoid: Day 42, n=18 | 2.7891 (145.0411)
  Norm CD20+/138+plasmacytoid: Day 56, n=19: number analyzed (Participants) | 19
  Norm CD20+/138+plasmacytoid: Day 56, n=19 | 20.1061 (220.7714)
  Norm CD20+/138+plasmacytoid: Day 84, n=19: number analyzed (Participants) | 19
  Norm CD20+/138+plasmacytoid: Day 84, n=19 | -44.0743 (65.0501)
  Norm CD20+/69+activated: Day 14, n=19: number analyzed (Participants) | 19
  Norm CD20+/69+activated: Day 14, n=19 | -0.9711 (196.9956)
  Norm CD20+/69+activated: Day 28, n=19: number analyzed (Participants) | 19
  Norm CD20+/69+activated: Day 28, n=19 | 106.5032 (379.9580)
  Norm CD20+/69+activated: Day 42, n=18: number analyzed (Participants) | 18
  Norm CD20+/69+activated: Day 42, n=18 | 9.8018 (138.7995)
  Norm CD20+/69+activated: Day 56, n=19: number analyzed (Participants) | 19
  Norm CD20+/69+activated: Day 56, n=19 | 15.6984 (132.7055)
  Norm CD20+/69+activated: Day 84, n=19: number analyzed (Participants) | 19
  Norm CD20+/69+activated: Day 84, n=19 | -18.3523 (120.1047)
  Norm CD20-/CD138+plasma cells: Day 14, n=20 | 24.3489 (151.0876)
  Norm CD20-/CD138+plasma cells: Day 28, n=20 | 21.4906 (180.2169)
  Norm CD20-/CD138+plasma cells: Day 42, n=19: number analyzed (Participants) | 19
  Norm CD20-/CD138+plasma cells: Day 42, n=19 | -6.6055 (129.1377)
  Norm CD20-/CD138+plasma cells: Day 56, n=20 | 3.0692 (175.5913)
  Norm CD20-/CD138+plasma cells: Day 84, n=20 | -51.0462 (38.0848)

ADVERSE EVENTS:
Time Frame: Up to Day 84
Description: Serious adverse events and non-serious adverse events were collected for the Safety Population which comprised of all the participants who received at least one dose of study medication.
Arm/Group | Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg (N=20)
Upper respiratory tract infection (Infections and infestations) | 4
Gingivitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Bone infarction (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Balanoposthitis (Reproductive system and breast disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02880852/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02880852/SAP_001.pdf